CLINICAL TRIAL: NCT04075929
Title: Aerobic Short or Long High Intensity Interval Training - Does it Matter
Brief Title: Short or Long High Intensity Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Responsible Party: Principal Investigator, Monica Klungland Torstveit, Professor, University of Agder
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Aerobic short og long interval
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Sports Performance; Cycling; Well-trained Athletes
Keywords: Cycling; endurance performance; intermittent exercise; maximal oxygen consumption; physiological adaptions; well-trained athletes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4x8 min (Other): 4x8-min intervals with 2-min recovery periods. The same accumulated duration of these three interval groups means that the total interval time is the same for each group: 4x8-min = 32 min
  Interventions: Other: Training effects on aerobic output
- 4x(8x40/20s) (Other): 4x(12x40/20-sec) intervals with 2-min recovery periods The same accumulated duration of these three interval groups means that the total interval time is the same for each group:4x(12x40/20-sec) = 32 min if the 20-sec recovery is not included in the total time of HIT
  Interventions: Other: Training effects on aerobic output
- 4x(12x40/20s) (Other): 4x(8x40/20-sec) intervals with 2-min recovery periods The same accumulated duration of these three interval groups means that the total interval time is the same for each group: 4x(8x40/20-sec) = 32 min if the 20-sec recovery is included in the total time of HIT
  Interventions: Other: Training effects on aerobic output

INTERVENTIONS:
Other: Training effects on aerobic output — The cyclists were allowed to perform ad libitum low intensity (LIT) in addition to high intensity (HIT) sessions that were determined to each group. The cyclists completed 12 supervised HIT sessions during the intervention period, three HIT sessions per week with at least 48 hours between each HIT-session. All HIT sessions were performed as supervised group training sessions. Each HIT session started with an individual 30 minutes' warm up at low intensity (55-70% HRmax) interspersed by freely chosen progressive sprints. For all groups the power output during the recovery periods was 50 % of the power output used during work intervals. The cyclists in all groups were instructed to perform each interval session at their maximal sustainable intensity. Each session ended with 15-20 minutes' cool down (55-70% HRmax). All HIT sessions were supervised and performed in groups on the University of Agder's (UiA) premises at Spicheren fitness center in Kristiansand.

SUMMARY:
To compare the effects of short and long high intensity interval training (HIT) conducted with the same total accumulated duration on physiological- and performance parameters during a 4-week training period.

DETAILED DESCRIPTION:
Studies among elite athletes have documented the importance of large amounts of training volume in order to perform at a high level in endurance sports. It is also well documented that both low intensity training (LIT), moderate intensity training (MIT) and high intensity training (HIT) should be included in the overall training efforts. It is well documented that HIT has a positive effect on the aerobic endurance among both elite athletes and recreational athletes.

Despite the fact that there is general agreement that HIT is an important part of the overall training, it is unclear how this part of the training should be organized in order to optimize the training effects. The adaptions of endurance performance seem to depend on both the intensity and the accumulated duration of the HIT sessions. Therefore, the aim of this study was to compare the effects of SI and LI training, including equal accumulated HIT duration, during a 4-week intervention period, conducted as 4x8-min with 2-min recovery periods, 4x(12x40/20-sec) with 2-min recovery periods and 4x(8x40/20-sec) with 2-min recovery periods, in different physiological- and performance parameters among well-trained cyclists.

ELIGIBILITY:
Inclusion Criteria:

* male < 40 years,
* peak oxygen uptake (VO2peak) > 55 ml.kg-1.min-1,
* training volume >3 sessions per week (within cycling)
* absence of disease and injuries.

Exclusion Criteria:

* disease/injuries
* frequent absence of HIT sessions during the period.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | 4 weeks
  VO2max

SECONDARY OUTCOMES:
Functional threshold power | 4 weeks
  FTP
Peak power output | 4 weeks
  PPO

CONTACTS AND LOCATIONS:
Overall Officials: Monica K. Torstveit, Professor, Principal Investigator — Universitetet i Agder
Locations (1):
- University of Agder, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: No